CLINICAL TRIAL: NCT00207922
Title: The Polarization and Expression of Chemokine Receptors of T Help Cell in the Pathogenesis of Acute and Chronic GVHD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Other Study IDs: DMR92-IRB-135
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2003-12

CONDITIONS: Hematopoietic Stem Cell Transplantation, Graft-Versus-Host Disease
Keywords: cytokine; T-cell; chemokine; graft-versus-host disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to see the correlation of polarization and the expresison of chemokine receptors of T help cells after allogeneic hematopoietic stem cell transplantation and clinical course graft-versus-host disease.

ELIGIBILITY:
Inclusion Criteria:

* patient received allogeneic stem cell transplantation at CMUH
* can be regularly followed at CMUH

Exclusion Criteria:

* patient who do not want to enter in this study

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Su-Peng Yeh, MD, Principal Investigator